CLINICAL TRIAL: NCT04116255
Title: Effects of Occlusal Splint and Therapeutic Home Exercises on Neuropathic Pain and Oral Health-related Quality of Life in Temporomandibular Disorders: a Randomized Prospective Study
Brief Title: Effects of Occlusal Splint and Therapeutic Home Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seçil Vural, Instructor of Physical Medicine and Rehabilitation,, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14719
Record Dates: First submitted 2019-09-30; First posted 2019-10-04 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Quality of Life; Neuropathic Pain; Somatic Pain
Keywords: Temporomandibular joint disorders; exercise therapy; occlusal splint; neuropathic pain
MeSH Terms: conditions — Neuralgia; Nociceptive Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: a randomized prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercises group (Experimental): exercises group apply regular therapeutic home exercises programme
  Interventions: Other: Temporomandibular joint Exercises
- splint group (Experimental): splint group use mandibular oral occlusal splint
  Interventions: Other: Mandibular oral occlusal splint

INTERVENTIONS:
Other: Mandibular oral occlusal splint — The panoramic open-mouth and close-mouth radiographs of the first group(splint group) were taken, and intraoral and extraoral examinations were performed by an experienced dentist that also examined the radiographs. The upper jaw of the patients was measured with an alginate impression material, to obtain a hard plaster model. Then, using these models, a vacuum plate machine made a customized mandibular oral occlusal splint suitable for each patient's teeth. The suitability of the splints was checked and confirmed by the dentist on the first and seventh days of use. The patients were asked to use these splints at night (for at least six hours) throughout the study.
  Arms: splint group
Other: Temporomandibular joint Exercises — This program was created by combining patient training and a home exercise program. The exercise program consisted of slow passive and active mouth opening and closing exercises, isometric masseter exercises, mouth stretching exercises, and resistant mouth opening and closing exercises. Each exercise set was administered twice a day, and each movement was undertaken for 10 seconds and repeated 15 times. The training was given by an experienced physical medicine and rehabilitation expert over approximately 45 minutes. The exercise program was demonstrated for the patients in front of a mirror, and each exercise was performed by a set of patients under the supervision of a doctor. A training document including the written exercise program was to the patients in the exercises group.
  Arms: exercises group

SUMMARY:
In this randomized controlled study, investigators planned to investigate the efficacy of oral occlusive splint and therapeutic home exercises in increasing the quality of life and reducing somatic and neuropathic pain in patients with temporomandibular joint dysfunction, determine their effects on other clinical data, and report long-term outcomes

DETAILED DESCRIPTION:
The aim of the present study to compare the efficacy of oral occlusive splint and therapeutic home exercises in increasing the quality of life and reducing somatic and neuropathic pain in patients with temporomandibular joint dysfunction and report long-term outcomes.

One hundred and one patients with temporomandibular joint dysfunction were included in the study. The patients were randomly divided into two groups: The first group received a mandibular oral occlusal splint and the second group was given a home exercise program for the temporomandibular joint. The patients were evaluated based on their maximum mouth opening, visual analog scale, short-form McGill pain questionnaire, painDETECT, oral health-related quality of health and hospital anxiety and depression scale scores at the beginning of treatment and at the end of the first and sixth months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of temporomandibular joint disorders for more than one month
* Being aged 18 to 60 years

Exclusion Criteria:

* History of trauma to temporomandibular joint or face
* History of an inflammatory joint disease
* Chronic analgesic use lasting more than six months
* Previous treatment for temporomandibular joint disorders
* History of a major psychiatric, neurological or neuromuscular disease (Lambert-Eaton syndrome, orofacial or tardive dyskinesia, myasthenia gravis)
* Migraine diagnosis
* Chronic headache or neck pain
* Chronic pain syndrome
* Pregnancy
* Disc displacement with or without reduction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Pain-free maximum mouth opening | six months
  This was measured in millimeters at the baseline and at each follow-up visit. The patients were asked to open their mouths as much as they could without having pain. Central incisors were measured in millimeters three times consecutively, and the highest measurement was recorded
Visual analog scale | six months
  The visual analogue scale is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. Ranges from 0 to 10 points, where the former indicates 'no pain' and the latter 'worst pain ever'. The patients were asked to mark the point that best represented the level of pain they experienced.
painDETECT | six months
  This scale is to evaluate the presence of neuropathic pain. PainDETECT incorporated an easy to use, patient- base questionnaire with nine items that do not require a clinical examination. There are seven weighted sensory descriptor items (''never'' to ''very strongly'') and two items relating to the spatial and temporal characteristics of the individual pain pattern. minimum score is 0 points and maximum score is 30 points. Patients with a total score of 12 or less are considered to have no neuropathic pain component. If the total score is between 13 and 18, it is assumed that a neuropathic component may be present although the result is not certain, and scores of 19 and above indicate the presence of a neuropathic pain component.
Oral health-related quality of health | six months
  This scale measures how an individual's oral health affects their quality of life and overall health, and how that they personally perceive this situation. A scoring known as oral health impact profile-14 is used, in which functional disability, physical pain, psychological disability, physical, psychological and social disability, and handicap measures are evaluated using two questions each. As the total score increases, the severity of the problem increases and the quality of life decreases.The minimum and maximum scores of this assessment tool is 0 and 56, respectively.

SECONDARY OUTCOMES:
Short-form McGill pain questionnaire | six months
  This is a multidimensional scale containing items that investigate the sensory and perceptual dimension of pain and examines the relationship between pain and anxiety, as well as pain intensity over time. The questionnaire is completed by patients.The main component of the short form McGill pain questionnaire consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1= mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. From this assessment scale, patients can score a minimum of 0 and a maximum of 112.

CONTACTS AND LOCATIONS:
Overall Officials: Secil Vural, Principal Investigator — Ankara Training and Research Hospital; Cagil Vural, Study Director — Ankara University, faculty of dentistry; Ali Ekemen, Principal Investigator — Ankara University, faculty of dentistry
Locations (1):
- Ankara Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No